CLINICAL TRIAL: NCT02296970
Title: An Observational Study to Determine the Clinical Cure Rate of Therapeutic up Front Shave Removal of Basal Cell Carcinoma of the Skin With Long Term Follow up to Evaluate Recurrence
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Timothy Patton, DO, Assistant Professor of Dermatology, University of Pittsburgh
Other Study IDs: PRO14020682
Record Dates: First submitted 2014-11-12; First posted 2014-11-21 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Deep shave removal using a blue surgical blade — Removal of a skin lesion with 2mm margins and an adequate amount of tissue deeper than the clinical appearance of the lesion using a blue surgical blade

SUMMARY:
Determine the effectiveness of a deep shave removal as a definitive treatment for basal cell carcinoma (BCC) without the need for a follow up surgical procedure.

DETAILED DESCRIPTION:
Basal cell carcinoma (BCC) is the most common skin cancer in the world, with approximately 3.5 million cases a year diagnosed in the United States. BCC are indolent and metastasis is extremely rare, occurring in less than .003% of cases. However, due to the high prevalence of this tumor, significant health care resources are used in its diagnosis and treatment. Management of BCC in many instances includes clinical evaluation of the lesion, biopsy or sampling of the lesion to confirm the diagnosis, followed by definitive treatment at a later date through surgical excision or medical therapy. A clinical diagnosis of BCC can be made with a high degree of confidence based on clinical findings. The investigators propose that by performing a deep shave removal of the entire lesion with histologically negative margins, based upon clinical diagnosis, complete removal can be achieved without the need for follow up therapy. Deep shave removal at time of initial evaluation is performed in many instances. The investigators believe that doing a deep shave removal would substantially reduce the number of second procedures that need to be done, thereby reducing treatment costs and patients' need to return for an additional procedure. In doing a deep shave removal, clinically diagnosed BCC will be removed entirely with narrow 2-3 mm margins, the tissue specimen will then be sent to the pathologist to confirm that margins are clear. The investigators will consider treatment of the BCC to be complete at this point and will follow the patients clinically.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older that are determined by an investigator to have a lesion that is highly likely to be a BCC, less than or equal to 1.0cm in largest diameter, based on clinical examination located in the trunk or extremities, proximal to the wrist and ankles
* Subject is able to give informed consent
* Subject is able to commit to 6 month follow up visit

Exclusion Criteria:

* BCC > 1cm in diameter on any one axis.
* Immunosuppressed patients
* Subjects with neutropenia
* Organ transplant patients
* Subjects with a life expectancy less than year
* Patients taking immunosuppressive medications, including prednisone at a dose of 10mg or greater with an expected duration greater than 4 weeks, azathioprine, mycophenolate mofetil, cyclosporine, oral Tacrolimus, any Tumor Necrosis Factor (TNF)-alpha inhibitor, ustekinumab, rituximab, or any other medication in the judgement of the investigator could results in clinically meaningful immunosuppression of the subject
* Basal cell carcinomas that have infiltrative or morpheaform characteristics based on clinical examination
* Subjects unable to provide informed consent
* Subjects unable to commit to 6 month follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 18 or older with the clinical diagnosis of BCC
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2014-12; Primary Completion 2016-06 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Measurement of clinical cure rate of deep shave removal in the treatment of BCC | 6 months

SECONDARY OUTCOMES:
Percentage of deep shave removal BCC with clear margins | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Patton, DO, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- Shadyside Place, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Ahnlide I, Bjellerup M. Accuracy of clinical skin tumour diagnosis in a dermatological setting. Acta Derm Venereol. 2013 May;93(3):305-8. doi: 10.2340/00015555-1560. PMID 23538779
- [Result] Ek EW, Giorlando F, Su SY, Dieu T. Clinical diagnosis of skin tumours: how good are we? ANZ J Surg. 2005 Jun;75(6):415-20. doi: 10.1111/j.1445-2197.2005.03394.x. PMID 15943729